CLINICAL TRIAL: NCT01338623
Title: Bioequivalence Study of Tansulosine 0,4 mg Capsule in Health Subjects -Fed State
Acronym: BET04cap
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Biocinese (Industry)
Responsible Party: Dr Josélia Larger Manfio, Biocinese
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: P03/11
Record Dates: First submitted 2011-04-18; First posted 2011-04-19 (Estimated); Last update posted 2011-05-03 (Estimated); Status verified 2011-04

CONDITIONS: Hyperplasia Prostatic
Keywords: bioequivalence; tansulosine
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tansulosine (Experimental)
  Interventions: Drug: Tansulosine

INTERVENTIONS:
Drug: Tansulosine — capsule 0,4 mg
  Other Names: Omics

SUMMARY:
The purpose of this study is to compare the bioavailability (rate and extent of absorption) of two tansulosine 0,4 mg capsule formulations. An open, randomized, two-period crossover study with a seven-days washout interval was conduced in 32 healthy male volunteers. The plasma samples were obtained up to 72 hours after drug administration. A sensitive and specific LC-MS/MS method was developed and validated for the determination of tansulosine in human plasma. Bioequivalence between the products was determined by calculating 90% confidence intervals for the ratio of Cmax, AUC 0-72h and AUC 0--inf.

DETAILED DESCRIPTION:
The study protocol was approved by Local Ethics Committee (UNICAMP - Campinas, Brazil). The study was performed with 32 healthy male volunteers. They were within 10% of their ideal body weight. Biochemical test and physical examination were carried out. Their medical history was also obtained. . Volunteers did not drink caffeine-containing drinks 48-hours before the study. The volunteers gave written informed consent to participate in study.

The study was designed as two-single-dose, randomized, open-label, balanced, crossover study, with two periods separated by 7-days washout. In both periods after a standard breakfast volunteers were given a single dose of their formulation (reference or test) of tansulosine with 200 mL of water. Blood samples (8 ml) were collected at 0 (pre-dose) and at 01:00; 02:00; 03:00; 04:00; 04;30; 05:00; 05:20; 05:40; 06:00; 06:20; 06:40; 07:00; 07:30; 08:00; 08:30; 09:00; 10:00; 12:00; 24:00; 48:00; 72:00h. These samples were centrifuged immediately and kept frozen at -20°C until the time of analysis. Standard meals were served at 4 and 8h after administration. During hospital confinement, volunteers were always under medical supervision.

ELIGIBILITY:
Inclusion Criteria:

* They were within 10% of their ideal body weight.
* Biochemical test and physical examination were carried out.
* No concomitant medications were allowed.
* Volunteers did not drink caffeine-containing drinks 48-hours before the study.
* The volunteers gave written informed consent to participate in the study.

Exclusion Criteria:

* Chronic disease
* Smokers

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2011-04; Primary Completion 2011-04 (Actual); Study Completion 2011-05 (Estimated)

PRIMARY OUTCOMES:
Bioequivalence interval | 3 months
  Bioequivalence between the products was determined by calculating 90% confidence intervals for the ratio of Cmax, AUC 0-72h and AUC 0--inf.

CONTACTS AND LOCATIONS:
Overall Officials: Josélia Manfio, Dr, Principal Investigator — Biocinese
Locations (1):
- Biocinese, Toledo, Paraná, Brazil